CLINICAL TRIAL: NCT03824847
Title: Immunomodulatory Effect of Macrolides in Naturally Occurring Influenza Virus Infections in the Community
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Community recruitment suspended due to COVID-19
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Dennis Kai-Ming Ip, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DKMI010.1
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Influenza, Human
Keywords: Macrolides; Immunomodulation
MeSH Terms: conditions — Influenza, Human | interventions — Clarithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Intervention group: clarithromycin 1 tablet (250mg) twice daily for three days
  Interventions: Drug: Clarithromycin 250 MG
- Placebo group (Placebo Comparator): Placebo group: (identical-looking) placebo 1 tablet twice daily for three days.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Clarithromycin 250 MG — Clarithromycin 1 tablet (250mg) twice daily for three days
  Arms: Intervention group
Drug: Placebos — Placebo group: (identical-looking) placebo 1 tablet twice daily for three days
  Arms: Placebo group

SUMMARY:
The investigators propose a double-blind randomised placebo-controlled study in naturally occurring influenza virus infections in the community setting to compare the impact of a short course of clarithromycin versus placebo, on the clinical course, viral shedding, immunomodulation, and the antimicrobial resistance pattern of respiratory bacterial carriage of the patients.

DETAILED DESCRIPTION:
Background: Influenza continues to pose an imminent threat to public health through seasonal epidemics and occasion pandemics with significant impact on morbidity and mortality. Increasing attention has also been paid in recent years to the potential benefit of immunomodulatory effect of macrolide antibiotics in the management of influenza virus infection.

Aims: To study the immunomodulatory effects of a short course of clarithromycin in naturally occurring influenza virus infection.

Design and subjects: The study is a double-blind, randomised controlled trial. One hundred adults aged 18-60 years will be recruited when they present with symptoms of acute respiratory infection within 48 hours of symptoms onset to university health clinics, and being tested positive with a QuickVue/Sofia (Quidel Corp., San Diego, CA) rapid influenza test. Consented patients tested positive with the rapid test will receive their clinical consultation and prescriptions as indicated as usual, and being randomised to receive either clarithromycin (250mg) or placebo (in a ratio of 1:1) taken twice daily orally for three days. Blood specimen, nasal and throat swabs will be collected on the same day (day 1). They will be followed-up on day 4, day 7 and day 10 for further collection of nasal and throat swabs, and serum samples. A symptom diary will be kept by each participant for 10 days for monitoring the clinical course of the infection.

Study instruments: QuickVue/Sofia (Quidel Corp., San Diego, CA) rapid influenza test, symptom diary, blood specimen, nasal and throat swabs.

Interventions: Intervention group: clarithromycin; placebo group: placebo in identical packaging.

Main outcome measures: The primary outcomes of the study will compare the duration of illness, viral shedding, patterns of plasma cytokine/chemokine and antimicrobial resistance pattern of respiratory bacterial carriage between patients who were randomised to clarithromycin or placebo.

Analysis: Intention to treat.

Potential significance: This will be the first placebo-controlled RCT to investigate the immunomodulatory effect of macrolide antibiotics in the management of influenza virus infection, in terms of its impact on the duration of illness, viral shedding, patterns of plasma cytokine/chemokine and antimicrobial resistance pattern of respiratory bacterial carriage. Findings from this study will have important contribution to our understanding on the potential immunomodulatory effect of macrolides, and help to inform the appropriate clinical management approach, and the potential

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18-60
* Presenting with symptoms of acute URTI (at least two among the following symptoms: body temperature ≥37.8°C, cough, rhinorrhea, sore throat, headache, myalgia/arthralgia) to university health clinics within 48 hours of illness onset.

Exclusion Criteria:

* Allergy to clarithromycin or any other macrolides or the ingredients in the tablets, which include microcrystalline cellulose, croscarmelose sodium, magnesium stearate and povidon will be excluded.
* Patients with a history of chronic liver disease, or any active lung, heart or renal diseases requiring regular medication, or any underlying immunocompromised condition or receiving immunosuppressive agents will also be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Time from recruitment to cessation of clinical illness | 10 days
  Defined as the time when all relevant clinical symptoms are resolved.
Time from recruitment to cessation of viral shedding | 10 days
  Defined as the time when no virus is detected by RT-PCR from both nasal and throat swabs.

SECONDARY OUTCOMES:
Duration and severity of individual symptoms | 10 days
  Participants will keep symptom diary twice daily for 10 days (from D1-D10), using 4-point scale of 0, 1, 2, or 3 for absent, mild, moderate, or severe symptoms respectively. Mild symptoms are easily tolerated and do not interfere with any usual activities; moderate symptoms interfere with usual activities; Severe symptoms are such that the individual cannot carry out usual activities. Ten common influenza symptoms (including feverishness, chills, cough, rhinorrhea, sore throat, general fatigue, headache, myalgia/arthralgia, vomiting, and diarrhea) will be recorded for ten days (D1-D10) and the duration of individual symptoms will be assessed.
Incidence of secondary complications | 28 days
  The symptom diary will be checked on each follow-up (D4, D7, and D10) and collected on D10 by our research staff when the patient returns for follow-up. Symptoms of possible side effects related to treatment (including skin rashes, nausea, vomiting, jaundice, dark urine) will be recorded. The occurrence of any complications including otitis media, bronchitis, sinusitis, and pneumonia will be enquired during all follow-up sessions and recorded, and cross checking with the attending doctor will be done where necessary.
Health-related quality of life | 28 days
  A simple quality of life (QOL) assessment based on two simple validated 11- point visual analog scales will also be done daily by all participants form D1 - D10, one to rate their own ability for performing normal daily activities (0 = unable to perform normal activity to 10 = fully able to perform normal activity) , and the other for a self-perceived overall health status over a 24-hour (0 = worst health to 10 = best possible health), both of which will be compared to an initial assessment of their normal pre-influenza state reported on the D1 baseline. All participants will also be required to complete the Acute Form of the Short Form-36, version 2 (SF-36), in D1, D10 and D28, for a more details assessment on the changes of Health-related quality of life (HRQL) related to the episode of the influenza infection.
Geometric mean rise in antibody titre against the infecting type or subtype of influenza virus | 28 days
  Paired sera will be collected on D1 and D28 for measuring the humoral antibody titres against the infecting type or subtype and other circulating strains of influenza viruses, and for evaluating the geometric mean titer rise from baseline to convalescence.
Changes in blood immunity (Cytokine/chemokine and pro-inflammatory mediators) | 7 days
  Plasma concentrations of 20+ cytokines/chemokines and proinflammatory mediators (e.g. IL-6, IL-8, TNFα, IFN-γ, IL-12p70 etc.) will be measured in each collected blood sample using cytokines bead assay by Flow cytometry.
Change in the carriage rate of common respiratory bacterial pathogen | 7 days
  change in the carriage rate of five common respiratory bacterial pathogen and the proportion of each that were macrolide resistant.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis KM Ip, MD, Principal Investigator — School of Public Health, The University of Hong Kong
Locations (1):
- School of Public Health, The University of Hong Kong, Hong Kong, Hong Kong